CLINICAL TRIAL: NCT04730115
Title: Evaluation of Architectural Changes in Mandibular Bone Pattern After Functional Treatment by Fractal Dimension Analysis
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, DİLARA NİL GÜNAÇAR, assistant professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2020/199
Record Dates: First submitted 2021-01-22; First posted 2021-01-29 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-01

CONDITIONS: Orthopedic Disorder
Keywords: Functional orthodontic appliances; fractal dimension; panoramic radiographs; orthodontics
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1. The treatment group (T): The treatment group comprised of 30 cases treated with functional appliance for one year in puberty.
- Group 2. The control group (C): The control group consists of 12 patients who had insufficient oral hygiene; didn't take any orthodontic treatment for one year.

SUMMARY:
In this study it was aimed to examine the changes in mandibular bone after functional treatment by using fractal dimension (FD) and cortical thickness (CT) analysis.

DETAILED DESCRIPTION:
In this study it was aimed to examine the changes in mandibular bone after functional treatment by using fractal dimension (FD) and cortical thickness (CT) analysis. The study will perform on 42 mandibular retrognathia cases. The treatment group (T), comprised of 30 cases treated with functional appliance for one year in puberty. The control group (C) consists of 12 patients who had insufficient oral hygiene; didn't take any orthodontic treatment for one year. FD and CT analysis will evaluate for both sides. FD measurements will perform on processus condylar, antigonial notch, and ramus regions in the panoramic radiographs. Paired t-test will apply to analyze all between groups (before (T1) and after treatment (T2), before (C1) and after (C2) control). Also, independent t-test wişll use to determine whether there was any difference between the treatment group (∆T=T2-T1) and the control group (∆C=C2-C1).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females were matched.
2. Treatment period of the treatment group was 1 year.
3. Observation period of the control group was also 1 year.
4. All groups had Class II malocclusion (ANB ≥ 5) with the retrognathic mandible in the period of puberty and had no systemic problem and impacted teeth.
5. Monoblock and twin-block appliances were applied to the treatment group.
6. Patients in the control group had insufficient oral hygiene and after oral-care was provided, they were taken into treatment.

Exclusion Criteriteria:

1. Radiographic images that do not have sufficient diagnostic quality

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The database was taken from the archives between 2017 and 2019 in Recep Tayyip Erdogan University. The study will consist of 30 cases treated with the functional appliance and 12 control patients who had insufficient oral hygiene were not treated for one year. After providing oral care cases were treated orthodontically.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
The effect of functional treatment on the cortical structure of the mandible will be investigated by measuring cortical thickness. | for one months from the beginning of the study
  the effects of functional treatment with cortical thickness to cortical bone structure
Thanks to fractal dimension analysis, the effect of functional treatment on the trabecular bone structure of the mandible will be examined. | for one week from the beginning of the study
  the effects of functional treatment with fractal analysis to trabecular bone structure

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Nil Günaçar, 1, Principal Investigator — Recep Tayyip Erdogan University Training and Research Hospital
Locations (1):
- Recep Tayyip Erdogan University Training and Research Hospital, Rize, Turkey (Türkiye)